CLINICAL TRIAL: NCT01265511
Title: A Phase 2a Study of SCY-635 in Combination With Peginterferon Alfa-2a (Pegasys) and Ribavirin (Copegus) in Treatment-Naive Subjects With Genotype 1 Hepatitis C Infection
Brief Title: Study of SCY-635, Pegasys and Copegus in Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCY-635-201
Record Dates: First submitted 2010-11-23; First posted 2010-12-23 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis C Infection
Keywords: Hepatitis C; SCY-635; Ribavirin; Interferon
MeSH Terms: conditions — Hepatitis C | interventions — SCY-635; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo + PegIFN + RBV for 4 weeks followed by PegIFN + RBV for 20 weeks
  Interventions: Drug: Placebo; Drug: Pegasys; Drug: Copegus
- SCY-635 600 mg (Active Comparator): SCY-635 600 mg + PegIFN + RBV for 4 weeks followed by PegIFN + RBV for 20 weeks
  Interventions: Drug: SCY-635; Drug: Pegasys; Drug: Copegus

INTERVENTIONS:
Drug: Placebo — Oral tablets given bid for 28 days
  Other Names: Batch # BMR/10/731
  Arms: Placebo
Drug: SCY-635 — SCY-635 tablets, 300 mg bid for 28 days
  Arms: SCY-635 600 mg
Drug: Pegasys — 180 ug prefilled syringe given once per week for up to 48 weeks
Drug: Copegus — tablets given bid for up to 48 weeks

SUMMARY:
This study will examine the effectiveness of 28 days of triple combination therapy including SCY-635 with peginterferon alfa 2a and ribavirin in reducing serum HCV RNA levels. An additional 20 weeks of treatment with the currently approved standard of care will be offered to all participants. The Week 24 visit will be the last on-study visit. After the Week 24 visit, all subjects with undetectable HCV RNA will be given the option to continue treatment with standard of care for an additional 24 weeks (out to Week 48) under the care of their Principal Investigator.

DETAILED DESCRIPTION:
Objectives:

The primary objective of this Phase 2a study was to assess the effect of treatment with SCY-635, used in combination with peginterferon alfa-2a (PegIFN α-2a) and ribavirin (RBV), on hepatitis C viral replication (as measured by quantitative serum HCV RNA) in treatment-naive subjects with chronic genotype 1 infection who have an IL28B genotype of C/T or T/T.

The secondary objective of the study was to evaluate the safety and pharmacokinetics (PK) of SCY-635 when given in combination with PegIFN α-2a and RBV.

Primary Endpoints:

Proportion of subjects in each cohort with an undetectable serum HCV RNA level at Week 4 of treatment

Secondary Endpoints:

Adverse events and clinical laboratory assessments, including tests of liver function Proportion of subjects achieving complete early virologic response (cEVR, defined as an undetectable serum HCV RNA level at Week 12) Proportion of subjects achieving partial early virologic response (pEVR, defined as a detectable serum HCV RNA level with ≥ 2 log10 reduction in serum HCV RNA from Baseline to Week 12) Proportion of subjects achieving an undetectable serum HCV RNA level at Week 24 Pharmacokinetic assessments of SCY-635 when given in combination with PegIFN α-2a and RBV; trough concentrations of PegIFN α-2a and RB

ELIGIBILITY:
Inclusion Criteria:

* Quantifiable serum levels of HCV-specific RNA in excess of 100,000 IU/mL
* Chronic HCV status
* HCV genotype 1 infection and IL28B genotype of C/T or T/T
* Liver biopsy results within 3 years prior to screening indicating the absence of cirrhosis

  *If no previous biopsy is available, a biopsy must be performed during the screening period to qualify for randomization
* Body mass index (BMI) between 18 and 38 kg/m2
* Laboratory variables within acceptable ranges:

  * ALT/AST < 3 × ULN;
  * HgB > 12g/dL for females, > 13 g/dL for males;
  * total WBC count > 3000/mm3 and ANC > 1500/mm3;
  * platelets > 100,000/mm3;
  * prothrombin time (or INR) ≤ 1.2 × ULN;
  * serum albumin ≥ 3.4 g/dL;
  * total bilirubin WNL;
  * serum creatinine WNL; if serum creatinine is > ULN, then calculated creatinine clearance must be > 100 mL/min (by Cockcroft-Gault formula) for subject to be eligible
* Subjects of childbearing potential (i.e., not surgically sterile or postmenopausal) must agree to use 2 forms of contraception from Screening until 24 weeks after completion of treatment with RBV
* Negative urine testing for amphetamines and cocaine at Screening.
* If female, the subject has a negative pregnancy test at Screening and on study Day 1

Exclusion Criteria:

* History of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease
* Females who are pregnant or breastfeeding
* Males with partners who are pregnant or are planning to become pregnant
* HCV genotype other than genotype 1 and an IL28B genotype of C/C
* Seropositive for HIV-1 or HIV-2 or hepatitis B virus (HBV) surface antigen (HBsAg)
* Use of any investigational agent within 3 months prior to dosing
* Received any prior FDA-approved or investigational drug or drug regimen for the treatment of hepatitis C
* Evidence of cirrhosis on a previous liver biopsy
* Evidence of decompensated liver disease
* Recipient of an organ transplant
* Evidence of hepatocellular carcinoma
* Evidence of ongoing alcohol or substance abuse
* Poorly-controlled diabetes mellitus
* Congestive heart failure or unstable cardiopulmonary condition, renal disease, or hemoglobinopathy (sickle cell anemia or thalassemia
* History of seizure disorder
* History of severe psychiatric illness, including severe depression, history of suicidal ideation, suicidal attempts, related hospitalizations, bipolar disorder, or psychosis requiring medication
* Concurrent medical condition or laboratory abnormality that would constitute a contra-indication for interferon use
* History of unstable thyroid disease that would preclude administration of interferon-based therapy
* Medical condition that requires use of systemic corticosteroids
* Received warfarin or other anticoagulants during the 21 days immediately prior to Screening, or is expected to require warfarin or other anticoagulants during the study.
* One or more additional known primary or secondary causes of liver disease, other than hepatitis C
* Any other concurrent medical condition likely to preclude compliance with the schedule of evaluations, or likely to confound the efficacy or safety observations
* 12-lead ECG showing the following:

  * Corrected QTc interval ≥ 450 msec (Bazett's correction);
  * QRS > 120 msec;
  * Clinically significant abnormalities;
* Severe retinopathy or other significant ophthalmological disorder
* Use of any herbal supplements within 28 days prior to dosing.
* The use of CYP3A inducers or inhibitors for at least 2 weeks prior to initiation of treatment through Week 6

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Muir, MD, Principal Investigator — Duke Clinical Research Institute; Keyur Patel, MD, Principal Investigator — Duke Clinical Ressearch Institute
Locations (4):
- United States (3):
  - Quest Clinical Research, San Francisco, California
  - Duke University Medical Center, Durham, North Carolina
  - Alamo Medical Research, San Antonio, Texas
- Fundacion de Investigation de Diego, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo + PegIFN + RBV for 4 weeks followed by PegIFN + RBV for 20 weeks
  Placebo: Oral tablets given bid for 28 days
  peginterferon alfa 2a: 180 ug prefilled syringe given once per week for up to 48 weeks
  Ribavirin: tablets given bid for up to 48 weeks
- SCY-635 600 mg: SCY-635 600 mg + PegIFN + RBV for 4 weeks followed by PegIFN + RBV for 20 weeks
  SCY-635: SCY-635 tablets, 300 mg bid for 28 days
  peginterferon alfa 2a: 180 ug prefilled syringe given once per week for up to 48 weeks
  Ribavirin: tablets given bid for up to 48 weeks
Period: Overall Study
Arm/Group | Placebo | SCY-635 600 mg
Started | 2 | 8
Completed | 0 | 5
Not Completed | 2 | 3
Not completed — Lack of Efficacy | 2 | 1
Not completed — Met stopping rules | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SCY-635 600 mg | Total
Number analyzed (Participants) | 2 | 8 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (15.56) | 44.6 (8.67) | 45.1 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 2 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 7 | 8
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 4 | 5
  Puerto Rico | 1 | 4 | 5
IL28B genotype [Number; unit: participants]
  IL28B_CT | 2 | 6 | 8
  IL28B_TT | 0 | 2 | 2
HCV genotype [Number; unit: participants]
  HCV_1a | 1 | 7 | 8
  HCV_1b | 1 | 1 | 2
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 7.21 (0.05) | 6.3 (0.49) | 6.48 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Undetectable HCV RNA
Time Frame: Week 4
Measure: Number; unit: participants
Arm/Group | Placebo | SCY-635 600 mg
Number analyzed (Participants) | 2 | 8
participants | 0 | 1

2. Secondary Outcome: Undetectable HCV RNA
Time Frame: Week 12
Measure: Number; unit: participants
Arm/Group | Placebo | SCY-635 600 mg
Number analyzed (Participants) | 2 | 8
participants | 0 | 3

3. Secondary Outcome: Partial Early Virologic Response
Description: Proportion of subjects with detectable HCV RNA that achieve a > or = 2 log reduction in HCV RNA from baseline to Week 12
Time Frame: Week 12
Measure: Number; unit: participants
Arm/Group | Placebo | SCY-635 600 mg
Number analyzed (Participants) | 2 | 8
participants | 0 | 4

4. Secondary Outcome: Undetectable HCV RNA
Time Frame: Week 24
Population: Week 24 analysis does not include the 2 placebo subjects because they were discontinued for lack of efficacy before week 24.
Measure: Number; unit: participants
Arm/Group | Placebo | SCY-635 600 mg
Number analyzed (Participants) | 0 | 8
participants |  | 5

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Placebo | SCY-635 600 mg
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/8
Other Adverse Events (participants affected / at risk) | 2/2 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2) | SCY-635 600 mg (N=8)
neutropenia (Blood and lymphatic system disorders) | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Fatigue (General disorders) | 1 | 2
Headache (Nervous system disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No